CLINICAL TRIAL: NCT04767984
Title: A Randomized and Placebo-Controlled Phase II Trial Targeting Dominant-Negative Missense Mutant P53 by Atorvastatin for Reducing the Risk of Longstanding Ulcerative Colitis-Associated Cancer
Brief Title: Testing Atorvastatin to Lower Colon Cancer Risk in Longstanding Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCI 20-02-02; P30CA060553 (NIH); UG1CA242643 (NIH); NCI-2021-01261 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI20-02-02 (Other: Northwestern University); NWU20-02-02 (Other: DCP)
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Carcinoma; Ulcerative Colitis
MeSH Terms: conditions — Colorectal Neoplasms; Colitis, Ulcerative | interventions — Atorvastatin; Colonoscopy; Biopsy; Specimen Handling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (atorvastatin, biospecimen collection) (Experimental): Patients receive atorvastatin PO QD for 12 months. Patients also undergo colonoscopy with biopsy, and collection of blood on the trial.
  Interventions: Drug: Atorvastatin Calcium; Procedure: Biopsy of Colon; Procedure: Biospecimen Collection; Other: Questionnaire Administration
- Arm II (placebo, biospecimen collection) (Placebo Comparator): Patients receive placebo PO QD for 12 months. Patients also undergo colonoscopy with biopsy, and collection of blood on the trial.
  Interventions: Procedure: Biopsy of Colon; Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Atorvastatin Calcium — Given PO
  Other Names: ATORVASTATIN CALCIUM TRIHYDRATE; CI-981; Lipitor
  Arms: Arm I (atorvastatin, biospecimen collection)
Procedure: Biopsy of Colon — Undergo colonoscopy with biopsy
  Other Names: Colonoscopic Biopsy; Colonoscopy and Biopsy
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo, biospecimen collection)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of atorvastatin in treating patients with ulcerative colitis who have a dominant-negative missense P53 mutation and are at risk of developing large intestinal cancer. Patients with ulcerative colitis are known to have an increased risk of developing large intestinal cancer. Better ways to control ulcerative colitis and more knowledge about how to prevent colon cancer are needed. Atorvastatin is a drug used to lower the amount of cholesterol in the blood and to prevent stroke, heart attack, and angina (chest pain). It blocks an enzyme that helps make cholesterol in the body. It also causes an increase in the breakdown of cholesterol. The information gained from this study may help doctors learn more about atorvastatin as an agent in cancer prevention, and may help to improve public health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of atorvastatin calcium (atorvastatin) treatment on reducing the fraction of colonic epithelial cells expressing mutant p53 protein detected via immunohistochemical staining in biopsy samples of colorectal mucosa obtained during colonoscopies done before and after atorvastatin intervention and compared to placebo control.

SECONDARY OBJECTIVES:

I. Examination of the effect of atorvastatin on the levels of biomarkers including Ki-67 (cell proliferation), Waf1p21 (wild type p53 allele reactivated signal), and cleaved caspase-3 (wild type p53-induced cell apoptosis) using immunohistochemistry (IHC) approach for colorectal biopsy specimens.

II. Examination of the effect of atorvastatin on the severity of histologic inflammation in colorectal biopsies using the Geboes grading system.

III. Examination of the effect of atorvastatin on the plasma concentration of cholesterol, high density lipoprotein (HDL) and low density lipoprotein (LDL) for monitoring atorvastatin effect on lowering cholesterol and its correlation with the levels of biomarkers in the colorectal biopsies.

IV. Examination of the effect of atorvastatin on the clinical efficacy on ulcerative colitis (UC) related symptoms using the Ulcerative Colitis Disease Activity Index (i.e. the Mayo score).

EXPLORATORY OBJECTIVES I. Examination of the effect of atorvastatin on the spectrum, hotspot and load of TP53 gene mutations using next generation sequencing and droplet digital polymerase chain reaction (PCR).

II. Will bank colorectal biopsies and blood samples and ribonucleic acid (RNA) and germline deoxyribonucleic acid (DNA) for future analyses, particularly on proteomics/prenylated protein profile, cytokine/chemokine profile, inflammatory lipid-mediator profile, RNA sequencing (RNAseq) and Chaperon/Co-chaperon proteins, etc.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive atorvastatin orally (PO) once daily (QD) for 12 months. Patients also undergo colonoscopy with biopsy, and collection of blood on the trial.

ARM II: Patients receive placebo PO QD for 12 months. Patients also undergo colonoscopy with biopsy, and collection of blood on the trial.

After completion of study treatment, patients are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have ulcerative colitis with > 8 years history and clinical remission (including the clinical remission for an extraintestinal manifestation/complication) confirmed by yearly surveillance endoscopy examination (Mayo grading < 3)
* They must be stable on maintenance therapy with mesalamine, thiopurines or biologics for over 3 months (Ulcerative Colitis Disease Activity Index [UCDAI] =< 1)
* A history of segmental colon resection is allowed
* UC in clinical remission, but with dysplasia-associated lesion or mass (DALM) at entry endoscope examination and DALM was completely resected by endoscopic mucosa resection, is allowed
* Participants 18-70 years old (both men and women). This is the standard age range for routine ulcerative colitis surveillance in adults
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* White blood cell count within normal institutional limits or absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits, unless known to have Gilberts syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (SGPT) =< 1.5 X institutional upper limit of normal (ULN)
* Creatinine =< 1.5 X institutional ULN
* Plasma level of cholesterol < 240 mg/dl or LDL-C < 190 mg/dl (since cholesterol > 240 mg/dl and LDL-C > 190 mg/dl need high dose (40 - 80 mg) atorvastatin per day to control hypercholesterolemia)
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Participants on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* Atorvastatin is contraindicated in pregnancy since it affects cholesterol synthesis pathway. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of baseline pregnancy test, throughout the duration of the study, and for 1 month following cessation of study drug. Females must begin adequate contraception immediately following screening pregnancy test. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately. If she is pregnant, she will be immediately withdrawn from the study and followed until the birth of the child
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Ulcerative proctitis (since patients with ulcerative proctitis have a significantly lower risk of developing colorectal cancer [CRC] than those with pancolitis or localized UC in left colon)
* Participants with medical conditions that, in the opinion of the investigator, would preclude the treatment intervention and colonoscopy, or limit ability to comply with therapy
* Participants with pancolitis or localized UC with total Mayo score >= 3 including Mayo endoscopic sub-score < 3 are excluded
* Use of corticosteroid therapy in the past 3 months due to high potential of relapse of active disease
* Use of statins in the last 12 months
* Use of any investigational drugs within the past 3 months
* A history of high-grade dysplasia or CRC or pan/severe colitis with total proctocolectomy
* History of chemotherapy within 2 years of screening
* History of allergic reactions attributed to atorvastatin
* Concomitant primary sclerosing cholangitis (PSC) with stage 4 liver fibrosis (biliary cirrhosis) and severe liver functional alteration
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding participants are excluded
* Human immunodeficiency virus (HIV)-positive participants are excluded due to anti-retroviral therapy that affect atorvastatin effect
* Children are excluded from this study since disease duration is usually < 8 years and there is no data about p53 mutation in this patient population
* Current use of cyclosporine, fibrates (e.g., gemfibrozil, fenofibrate), strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, posaconazole, voriconazole, human immunodeficiency virus (HIV) protease inhibitors, boceprevir, telaprevir, erythromycin, clarithromycin, telithromycin, nefazodone, or cobicistat-containing products), or strong CYP3A4 inducers (e.g., carbamazepine, phenytoin, rifampin, St. John's wort, bosentan, efavirenz, etravirine, modafinil, nafcillin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in mutant p53 staining in biopsy samples obtained during colonoscopies done before and after intervention | Up to 2 years
  Counted as p53 positive cells/100 epithelial cells under at least 5 high powered fields per slide or 100 crypts or 2000 cells/slide per biopsy, measured by immunohistochemistry (IHC) staining. The level of biomarker expression will be determined by chromogenic staining. Because multiple samples will be obtained per participant, participant-level %p53 mutation will be summarized as the average %p53 across these samples. Descriptive statistics will be used to summarize changes in each arm, as well as the difference in change between arms. Analysis will be conducted using a two-sample t-test comparing within-subject changes in average percentage (%) p53 between treatment arms. A more comprehensive analysis will be done using a linear mixed effects model, where the outcome variable will be %p53 staining in each sample evaluated at baseline and post-treatment.

SECONDARY OUTCOMES:
Levels of biomarkers of Ki-67 (cell proliferation), Waf1p21 (wild type p53 allele reactivated signal), and cleaved caspase-3 (wild type p53-induced cell apoptosis) | Up to 2 years
  Using IHC approach for colorectal biopsy specimens.
Histological analysis for grading the severity of histologic inflammation in colorectal biopsies | Up to 2 years
  Using the Geboes grading system (grading score: 0 - 4). Highest grade histology and extent of UC (pancolitis vs localized UC) across multiple samples will be used at each time point. Changes in scores from baseline to post-treatment will be calculated, and compared between arms using the Wilcoxon rank sum test.
Plasma concentration of cholesterol, high density lipoprotein (HDL) and low density lipoprotein (LDL) | Up to 2 years
  Will monitor atorvastatin effect on lowering cholesterol and its correlation with the levels of biomarkers in the colorectal biopsies. Changes in plasma concentration of cholesterol, HDL and LDL (for monitoring atorvastatin effect on lowering cholesterol) will be compared between treatment arms using similar approaches as the primary analysis of %TP53 described above. The association of plasma concentration of cholesterol, HDL and LDL with the levels of biomarkers in the colorectal biopsies will be analyzed using linear mixed models as described above with plasma level added to the model as a fixed effect. Separate models will be fitted for each type of cholesterol (total, HDL and LDL).
Clinical efficacy on UC related symptoms | Up to 2 years
  Using the Ulcerative Colitis Disease Activity Index (activity score: 0 - 4) (i.e. the Mayo score).

OTHER OUTCOMES:
Analysis of spectrum, hotspot and load of TP53 gene mutations | Up to 2 years
  Using next generation sequencing and droplet digital polymerase chain reaction (PCR) technologies. The spectrum of TP53 mutations will be analyzed for frequency of each hotspot mutation in each group. For analyzing binary variables (presence or absence of each hot spot mutation), a Pearson's chi-squared test will be used. Frequency of each hotspot mutation for each noted group will be provided as descriptive measures of location and variance. The load of TP53 mutations in the biopsy specimens will be quantified as the ratio of mutant allele to wild-type allele using droplet digital PCR and allele-specific primers. Descriptive statistics will be used to summarize these at each time point for each treatment arm. Changes in TP53 mutation load, a continuous biomarker, will be compared between treatment arms using similar approaches as the primary analysis of %TP53 described above.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Hanauer, MD, Study Chair — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://sharing.nih.gov/